CLINICAL TRIAL: NCT05147376
Title: Effectiveness of a Curcumin Mouthwash in Preventing Traumatic Ulcers in Patients With Fixed Orthodontic Appliances: a Randomized Clinical Trial
Brief Title: Effectiveness of a Curcumin Mouthwash in Preventing Traumatic Ulcers in Patients With Fixed Orthodontic Appliances
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Supaporn Suttamanatwong, D.D.S., Ph.D, Department of Physiology, Faculty of Dentistry, Chulalongkorn University, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HREC-DCU 2021-044
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Oral Ulcer; Orthodontic Appliances, Fixed
Keywords: Curcumin; Curcumin mouthwash; Traumatic ulcers; Fixed orthodontic appliances
MeSH Terms: conditions — Oral Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This clinical trial is a double-blind study that participants and examiner will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumin mouthwash (Experimental): The curcumin mouthwash contains the final concentration of 1 μM curcumin, water, xylitol, and food coloring agent.
  Interventions: Drug: Curcumin mouthwash
- Placebo mouthwash (Sham Comparator): The placebo mouthwash contains water, xylitol, and food coloring agent.
  Interventions: Drug: Placebo mouthwash

INTERVENTIONS:
Drug: Curcumin mouthwash — Rinse with 10 ml for 1 minute, twice a day for 28 days after brushing in the morning and at night, following proper oral hygiene and avoid taking any liquid or food for 30 minutes after rinsing.
  Arms: Curcumin mouthwash
Drug: Placebo mouthwash — Rinse with 10 ml for 1 minute, twice a day for 28 days after brushing in the morning and at night, following proper oral hygiene and avoid taking any liquid or food for 30 minutes after rinsing.
  Arms: Placebo mouthwash

SUMMARY:
The study is a randomized controlled trial. The participants will be equally allocated into 2 groups to compare clinical effectiveness of curcumin mouthwash in fixed orthodontic patients during the first month of treatment.

DETAILED DESCRIPTION:
Patients who require fixed orthodontic appliances as part of their orthodontic treatment at the Faculty of Dentistry, Chulalongkorn University will be asked if they will volunteer for this clinical research. Participants will be informed about the objectives of the study, study process, advantages, disadvantages before making a decision to participate in this study. The consent form will be signed prior to participating in the study. A week before bracket cementation visit, a participant will attend his/her appointment for a full clinical history taking and oral screening exam by one examiner. Each participant will be allocated by a trial number and receive 3 bottles of either placebo or curcumin mouthwash accordingly. A tube of sodium lauryl sulfate (SLS)-free, non-herbal toothpaste and 1 toothbrush will be provided to each participant. Moreover, the instruction VDO will be given to participants to "Rinse with 10 ml for 1 minute, twice a day for 28 days after brushing in the morning and at night, following proper oral hygiene and avoid taking any liquid or food for 30 minutes after rinsing" in the first 28 days after bracket cementation. Then, participants will be provided with a daily record form on Google Form and requested to record every day during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Fixed orthodontic patients aged 12-30 years old
* Fixed orthodontic appliances on at least 1 arch (at least 10 teeth per arch)
* Patients with good general health without any systemic diseases
* Patients who are not using any herbal toothpaste or any mouthwash in daily life for the past 2 weeks
* Patients who are not taking any medications which may influenced the pattern of oral ulceration
* Patients who are willing and able to cooperate with all aspects of the protocol and able to communicate effectively and give informed written consent from parents if patients are younger than 18 years old

Exclusion Criteria:

* Cigarette smoking
* History of hypersensitivity or allergy to turmeric or other ingredients of mouthwash
* History of oral mucosal lesions and skin diseases
* Oral ulceration or inflammation with unknown etiology
* Pregnant or lactating women

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Incidence of traumatic ulcer | 28 days
  The question in Google Form will ask about the number of traumatic ulcers that can be obviously seen in the mouth. The examiner will provide a picture of traumatic ulcer in the first visit. The participant will be requested to closely check on their mouth starting from reversing the upper and lower lips, then inspect the inner surface of lip and gingiva. Second, move buccal mucosa away from the teeth and gingiva, then, examine one side to the other. The participant will be requested to mark the site of traumatic ulcers on the simple diagram of oral cavity which is divided into 6 area per arch (Right molar teeth, right premolar teeth, right anterior teeth, left molar teeth, left premolar teeth, left anterior teeth). The incidence will be recorded dichotomously (presence or absence of traumatic ulcers).
Duration of each ulcer until it heals | 28 days
  A period between the first day that traumatic ulcer can be seen unit it resolves. As the participant will be requested to record number of ulcers and locate the sites every day. Duration will be calculated at the end of trial

SECONDARY OUTCOMES:
Pain score | 28 days
  The pain score will be evaluated by participant based on visual analog scale . The participant will be asked to select a number on the scale that describe the most of their pain and record the state number between 0-100. A higher score represents greater pain intensity
The site of traumatic ulcer | 28 days
  The participants will be requested to mark the site of any ulcer on simple diagram of oral cavity which is represented by a number on each of the divided 6 area of buccal mucosa per arch, the most common area of traumatic ulcer (Right molar teeth, right premolar teeth, right anterior teeth, left molar teeth, left premolar teeth, left anterior teeth).
Use of orthodontic wax | 28 days
  The participants will be asked to mark the site of using orthodontic wax on a simple diagram of oral cavity which is represented by a number on each of the divided 6 area per arch (Right molar teeth, right premolar teeth, right anterior teeth, left molar teeth, left premolar teeth, left anterior teeth).
Comments of adverse effect (if any) | 28 days
  The participants will be asked to record in Google Form daily for any complaint of discomfort from using mouthwash.
Comments of participant's satisfaction | 28 days
  At the end of the clinical trial, the participants will be asked to record for levels of satisfaction in mouthwash. The score will be numbered from very satisfied at score 5, satisfied at score 4, neutral or OK at score 3, dissatisfied at score 2, and very dissatisfied at score 1.
Comments of any suggestions | 28 days
  At the end of the clinical trial, the participants will be asked to record for any suggestions and comments about the trial or mouthwash.

CONTACTS AND LOCATIONS:
Overall Officials: Supaporn Suttamanatwong, D.D.S.,Ph.D., Principal Investigator — Department of Physiology, Faculty of Dentistry, Chulalongkorn University
Locations (1):
- Department of Pediatric Dentistry, Postgraduate dental clinic, Faculty of Dentistry, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akbik D, Ghadiri M, Chrzanowski W, Rohanizadeh R. Curcumin as a wound healing agent. Life Sci. 2014 Oct 22;116(1):1-7. doi: 10.1016/j.lfs.2014.08.016. Epub 2014 Sep 6. PMID 25200875
- [Background] Baricevic M, Mravak-Stipetic M, Majstorovic M, Baranovic M, Baricevic D, Loncar B. Oral mucosal lesions during orthodontic treatment. Int J Paediatr Dent. 2011 Mar;21(2):96-102. doi: 10.1111/j.1365-263X.2010.01078.x. Epub 2010 Dec 2. PMID 21121986
- [Background] Chattopadhyay I, Biswas K, Bandyopadhyay U, Banerjee RK. Turmeric and curcumin: Biological actions and medicinal applications. CURRENT SCIENCE-BANGALORE-. 2004;87:44-53.
- [Background] Duggi S, Handral H, Handral R, G T, Sd DS. Turmeric: Nature's precious medicine. Asian Journal of Pharmaceutical and Clinical Research. 2013;6:10-6.
- [Background] Emiroglu G, Ozergin Coskun Z, Kalkan Y, Celebi Erdivanli O, Tumkaya L, Terzi S, Ozgur A, Demirci M, Dursun E. The Effects of Curcumin on Wound Healing in a Rat Model of Nasal Mucosal Trauma. Evid Based Complement Alternat Med. 2017;2017:9452392. doi: 10.1155/2017/9452392. Epub 2017 Sep 5. PMID 29018487
- [Background] Fitzpatrick SG, Cohen DM, Clark AN. Ulcerated Lesions of the Oral Mucosa: Clinical and Histologic Review. Head Neck Pathol. 2019 Mar;13(1):91-102. doi: 10.1007/s12105-018-0981-8. Epub 2019 Mar 7. PMID 30701449
- [Background] Jurenka JS. Anti-inflammatory properties of curcumin, a major constituent of Curcuma longa: a review of preclinical and clinical research. Altern Med Rev. 2009 Jun;14(2):141-53. PMID 19594223
- [Background] Khan RMS, Hassan KR, Rizwan M, Ashraf J. Prevalence and type of oral mucosal lesions in patients with fixed orthodontic appliances. Medical Forum Monthly. 2016;27:12-5.
- [Background] Lau P, Wong R, editors. Risks and complications in orthodontic treatment, 2006.
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Mahattanadul S, Mustafa MW, Kuadkaew S, Pattharachayakul S, Ungphaiboon S, Sawanyawisuth K. Oral ulcer healing and anti-Candida efficacy of an alcohol-free chitosan-curcumin mouthwash. Eur Rev Med Pharmacol Sci. 2018 Oct;22(20):7020-7023. doi: 10.26355/eurrev_201810_16173. PMID 30402869
- [Background] McHugh ML. Interrater reliability: the kappa statistic. Biochem Med (Zagreb). 2012;22(3):276-82. PMID 23092060
- [Background] Mohanty C, Sahoo SK. Curcumin and its topical formulations for wound healing applications. Drug Discov Today. 2017 Oct;22(10):1582-1592. doi: 10.1016/j.drudis.2017.07.001. Epub 2017 Jul 12. PMID 28711364
- [Background] Mondal S, Ghosh S, Moulik SP. Stability of curcumin in different solvent and solution media: UV-visible and steady-state fluorescence spectral study. J Photochem Photobiol B. 2016 May;158:212-8. doi: 10.1016/j.jphotobiol.2016.03.004. Epub 2016 Mar 6. PMID 26985735
- [Background] Nagpal M, Sood S. Role of curcumin in systemic and oral health: An overview. J Nat Sci Biol Med. 2013 Jan;4(1):3-7. doi: 10.4103/0976-9668.107253. PMID 23633828
- [Background] Neville BW, Damm DD, Allen CM, Chi AC. Physical and Chemical Injuries. In: Oral & Maxillofacial Pathology. 4th ed. Elsevier: Missouri; 2016. p. 259-309.
- [Background] Noble J. Managing pain or discomfort caused by orthodontic appliances. J Can Dent Assoc. 2013;79:d45. No abstract available. PMID 23763732
- [Background] Rebelo MAB, Correra de Queiroz A. Gingival Indices: State of Art, Gingival Diseases-Their Aetiology, Prevention and Treatment. Publisher: InTech. 2011:41-2.
- [Background] Rujirachotiwat A, Suttamanatwong S. Curcumin Promotes Collagen Type I, Keratinocyte Growth Factor-1, and Epidermal Growth Factor Receptor Expressions in the In Vitro Wound Healing Model of Human Gingival Fibroblasts. Eur J Dent. 2021 Feb;15(1):63-70. doi: 10.1055/s-0040-1715781. Epub 2020 Oct 1. PMID 33003239
- [Background] Rujirachotiwat A and Suttamanatwong S. Effect of Curcuminonthe Expression of Wound Healing-related Genes in Human Gingival Fibroblasts.
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMC Med. 2010 Mar 24;8:18. doi: 10.1186/1741-7015-8-18. PMID 20334633
- [Background] Shamash MSA, Zaidan TF. Effect of topical curcumin on the healing of major oral mucosal ulceration. EurAsian Journal of BioSciences. 2020;14:4653-60.
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] Smith PC, Martínez C. Wound Healing in the Oral Mucosa. In: Bergmeier LA, editor. In: Oral Mucosa in Health and Disease: A Concise Handbook. Cham: Springer International Publishing; 2018. p. 77-90.
- [Background] Soleimani V, Sahebkar A, Hosseinzadeh H. Turmeric (Curcuma longa) and its major constituent (curcumin) as nontoxic and safe substances: Review. Phytother Res. 2018 Jun;32(6):985-995. doi: 10.1002/ptr.6054. Epub 2018 Feb 26. PMID 29480523
- [Background] Travess H, Roberts-Harry D, Sandy J. Orthodontics. Part 6: Risks in orthodontic treatment. Br Dent J. 2004 Jan 24;196(2):71-7. doi: 10.1038/sj.bdj.4810891. PMID 14739957
- [Background] Zaher A, Elsabaa H, Abou Elkhier M, Elhindawy M. Impact of curcumin on tongue ulcer healing in albino rats. Mansoura J Dent. 2014;1:85-9.
- [Result] Akbari G, Setiani T, Malik I. Traumatic ulcer distribution of patiens with removable orthodontic appliance in Orthodontics Clinics of Dental Specialist Program. Padjadjaran Journal of Dentistry. 2014;26
- [Result] Al-Maweri SA, Alaizari N, Alharbi AA, Alotaibi SA, AlQuhal A, Almutairi BF, Alhuthaly S, Almutairi AM. Efficacy of curcumin for recurrent aphthous stomatitis: a systematic review. J Dermatolog Treat. 2022 May;33(3):1225-1230. doi: 10.1080/09546634.2020.1819529. Epub 2020 Sep 9. PMID 32893718
- [Result] Asher C, Shaw WC. Benzydamine hydrochloride in the treatment of ulceration associated with recently placed fixed orthodontic appliances. Eur J Orthod. 1986 Feb;8(1):61-4. doi: 10.1093/ejo/8.1.61. No abstract available. PMID 3514243
- [Result] Deshmukh RA, Bagewadi AS. Comparison of effectiveness of curcumin with triamcinolone acetonide in the gel form in treatment of minor recurrent aphthous stomatitis: A randomized clinical trial. Int J Pharm Investig. 2014 Jul;4(3):138-41. doi: 10.4103/2230-973X.138346. PMID 25126527
- [Result] Kluemper GT, Hiser DG, Rayens MK, Jay MJ. Efficacy of a wax containing benzocaine in the relief of oral mucosal pain caused by orthodontic appliances. Am J Orthod Dentofacial Orthop. 2002 Oct;122(4):359-65. doi: 10.1067/mod.2002.126405. PMID 12411880
- [Result] Kvam E, Bondevik O, Gjerdet NR. Traumatic ulcers and pain in adults during orthodontic treatment. Community Dent Oral Epidemiol. 1989 Jun;17(3):154-7. doi: 10.1111/j.1600-0528.1989.tb00012.x. PMID 2736897
- [Result] Kvam E, Gjerdet NR, Bondevik O. Traumatic ulcers and pain during orthodontic treatment. Community Dent Oral Epidemiol. 1987 Apr;15(2):104-7. doi: 10.1111/j.1600-0528.1987.tb00493.x. PMID 3471374
- [Result] Leiva-Cala C, Lorenzo-Pouso AI, Centenera-Centenera B, Lopez-Palafox J, Gandara-Vila P, Garcia-Garcia A, Perez-Sayans M. Clinical efficacy of an Aloe Vera gel versus a 0.12% chlorhexidine gel in preventing traumatic ulcers in patients with fixed orthodontic appliances: a double-blind randomized clinical trial. Odontology. 2020 Jul;108(3):470-478. doi: 10.1007/s10266-019-00468-w. Epub 2019 Oct 29. PMID 31664632
- [Result] Mainali A. Occurrence of Oral Ulcerations in Patients undergoing Orthodontic Treatment: A Comparative study. Orthodontic Journal of Nepal. 2014;3.
- [Result] Manifar S, Obwaller A, Gharehgozloo A, Boorboor Shirazi Kordi H, Akhondzadeh S. Curcumin Gel in the Treatment of Minor Aphthous Ulcer: a Randomized, Placebo- Controlled Trial. J Med Plants. 2012;11(41):40-5.
- [Result] Patil K, Guledgud MV, Kulkarni PK, Keshari D, Tayal S. Use of Curcumin Mouthrinse in Radio-Chemotherapy Induced Oral Mucositis Patients: A Pilot Study. J Clin Diagn Res. 2015 Aug;9(8):ZC59-62. doi: 10.7860/JCDR/2015/13034.6345. Epub 2015 Aug 1. PMID 26436049
- [Result] Rennick LA, Campbell PM, Naidu A, Taylor RW, Buschang PH. Effectiveness of a novel topical powder on the treatment of traumatic oral ulcers in orthodontic patients: A randomized controlled trial. Angle Orthod. 2016 May;86(3):351-7. doi: 10.2319/050415-303.1. Epub 2015 Sep 24. PMID 26401826
- [Result] Sharma RA, Euden SA, Platton SL, Cooke DN, Shafayat A, Hewitt HR, Marczylo TH, Morgan B, Hemingway D, Plummer SM, Pirmohamed M, Gescher AJ, Steward WP. Phase I clinical trial of oral curcumin: biomarkers of systemic activity and compliance. Clin Cancer Res. 2004 Oct 15;10(20):6847-54. doi: 10.1158/1078-0432.CCR-04-0744. PMID 15501961
- [Result] Shaw WC, Addy M, Griffiths S, Price C. Chlorhexidine and traumatic ulcers in orthodontic patients. Eur J Orthod. 1984 May;6(2):137-40. doi: 10.1093/ejo/6.2.137. No abstract available. PMID 6587971
- [Result] Waghmare PF, Chaudhari AU, Karhadkar VM, Jamkhande AS. Comparative evaluation of turmeric and chlorhexidine gluconate mouthwash in prevention of plaque formation and gingivitis: a clinical and microbiological study. J Contemp Dent Pract. 2011 Jul 1;12(4):221-4. doi: 10.5005/jp-journals-10024-1038. PMID 22186854
- [Derived] Somprajob C, Auychai P, Chavanavesh J, Suttamanatwong S. Effectiveness of curcumin mouthwash in preventing traumatic ulcers in orthodontic patients. BMC Oral Health. 2025 Nov 3;25(1):1725. doi: 10.1186/s12903-025-07141-5. PMID 41185016